CLINICAL TRIAL: NCT07089095
Title: Factors and Preferences in Patient Selection of Rehabilitation Care Following Acute Stroke
Brief Title: Factors and Preferences in Patient Selection of Rehabilitation Care Following Acute Stroke: A Predictive Correlational Study.
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202302129RIND
Record Dates: First submitted 2023-06-04; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-04

CONDITIONS: Acute Stroke
Keywords: patient preferences
MeSH Terms: conditions — Stroke; Patient Preference | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- acute stroke patient: If acute stroke patient test on the Short Portable Mental State Questionnaire, assessment results are cognitively complete (0-2 questions wrong) or mild (3-4 questions wrong) cognitive impairment, and the patients participate in the study with informed consent.
  Interventions: Other: questionnaire
- acute stroke family: Family members of those with acute stroke patients are moderate (5-7 wrong answers) or severe (8-10 wrong answers) cognitive impairments assessed by the Short Portable Mental State Questionnaire (SPMSQ) participated in the study with informed consent.
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — This is a Relation Research. Use the patient decision aids for acute stroke rehabilitation, then data are collected with patients' characteristics, National Institutes of Health Stroke Scale (NIHSS), Barthel Index (BI), Modified Rankin Scale (mRS), and factors and preferences in the patient selection of rehabilitation care questionnaire.

SUMMARY:
Background and Purpose Patients with stroke have to receive the rehabilitation care after medical condition has stabilized. In recent years, the long-term care policy offers more options available for rehabilitation care after stroke. However, the selection of care is mainly based on physcicians' advice. This study explores the factors and preferences in patient selection of rehabilitation care following acute stroke, in order to help clinical health professionals incorporate patients' preferences in patient-centred care to properly arrange the stroke rehabilitation care.

Methods This is a cross-sectional and predictive study. Purposive sampling of patients surviving acute stroke is taken in the general ward of a medical center in northern Taiwan. Data are collected with patients' characteristics, National Institutes of Health Stroke Scale (NIHSS), Barthel Index (BI), Modified Rankin Scale (mRS), and factors and preferences in patient selection of rehabilitation care questionnaire. Data are analyzed using IBM SPSS 26.0 for windows. Demographic and clinical characteristics, family support systems and health care systems are compared between patients' preference in the selections of rehabilitation care. Variables with p < .05 are included as potential predictor variables in the subsequent logistic regression analysis. The level of statistical significance is set at α=0.05.

Expected results Demographic and clinical characteristics, family support systems and health care systems are expected as potential predictors of patients' preference in the selection of rehabilitation care.

ELIGIBILITY:
Inclusion Criteria:

* Age≧18 years old.
* Patients with stroke (International Classification of Disease, ICD 10th edition I60-I68, G45-G46) diagnosed by physicians within 2 weeks after the onset of stroke, including the first and second strokes.

Exclusion Criteria:

* Those with a score of 5 on the Modified Rankin Scale (mRS).
* Those who have been accepted as research subjects have been admitted to hospital again for stroke.
* People living in rehabilitation wards.
* Those with unstable vital signs.
* Those receiving palliative care or care.
* Patients or family members who cannot communicate in Chinese or Taiwanese.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stroke (International Classification of Disease, ICD 10th edition I60-I68, G45-G46)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2025-07-25 (Estimated); Study Completion 2025-07-25 (Estimated)

PRIMARY OUTCOMES:
Patient preferences questionnaire | 2025/1/31
  Patient preferences include：post-acute care, inpatient rehabilitation, outpatientrehabilitation, reablement at home.

SECONDARY OUTCOMES:
Patients' characteristics | 2025/1/31
  Questionnaire include:gender, age, comorbidities, indwelling line, stroke type, day-onset stroke, times of stroke, pre-stroke functional level.
Stroke severity | 2025/1/31
  National Institutes of Health Stroke Scale (NIHSS) The NIHSS score ranges from 0 to 42,with higher scores indicating greater severity of stroke symptoms.
Activities of Daily Living | 2025/1/31
  Barthel Index (BI) It refers to the following 10 categories: feeding, bathing, grooming, dressing, bowel control, bladder control, toileting, chair transfer, ambulation and stair climbing. Items are weighted according to the level of nursing care required and are rated in terms of whether individuals can perform activities independently, with some assistance, or are dependent (scored as 10, 5 or 0).
Level of post-stroke functional independence | 2025/1/31
  Modified Rankin Scale (mRS). It consisted of a single item, with five grades representing no, slight, moderate, moderately severe, and severe disability.
Factors and preferences in patient selection of rehabilitation | 2025/1/31
  Questionnaire include:
social circumstances | 2025/01/31
  Questionnaire include:

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No